CLINICAL TRIAL: NCT05618652
Title: Development and Pilot Testing of an Equity-focused and Trauma-informed Communication Intervention During Family-centered Rounds
Brief Title: Pilot Testing of an Equity Focused and Trauma-informed Communication Intervention During Family-centered Rounds
Acronym: EFTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00111356; 1K23MD018433 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-11-16 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hospitalism in Children; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The investigators will test the intervention in a randomized pilot with intervention and waitlist control arms. Half the clinical teams will receive the clinician communication intervention immediately upon enrollment and half will receive the intervention after 6 months. The investigators will assess recruitment, enrollment, and data collection feasibility as well as intervention fidelity to evaluate feasibility of implementation and skill uptake using audio-recordings of rounds. The investigators will develop a semi-structured interview and survey to assess acceptability as well as facilitators/barriers to implementation.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and their caregivers will not know whether their clinical team has received or not yet received the communication intervention. Additionally, team members who assess outcomes (coding of audio-recorded transcripts) will be blinded to the clinical team intervention status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician Coaching Immediate Intervention Arm-- Caregivers (Active Comparator): Clinicians who receive the intervention will participate for up to 12 months, which includes completion of didactics, 8 audio-recorded clinical encounters, 4 feedback sessions, and completion of a post-intervention brief interview and survey. After completing didactic training elements, clinicians will receive coaching and professional feedback on their communication with caregivers of children in the hospital. The investigators will provide clinicians with illustrative examples from their encounters to prompt discussion and self-reflection.
  Caregivers of hospitalized children will not know if their clinician has received the communication intervention. The investigators will recruit 40 caregivers in this arm.
  Interventions: Behavioral: Equity Focused and Trauma-Informed Communication Intervention
- Clinician Coaching Wait-List Control Arm-- Caregivers (Other): Clinicians in the wait-list control arm will initially serve as the control arm then receive the intervention to provide feasibility and acceptability data. The clinicians randomized the control arm will undergo didactics and feedback once their pre-intervention audio-recordings are complete.
  Caregivers of hospitalized children will not know if their clinician has yet received the communication intervention. The investigators will recruit 40 caregivers in this arm prior to clinicians receiving the intervention.
  Interventions: Behavioral: Equity Focused and Trauma-Informed Communication Intervention

INTERVENTIONS:
Behavioral: Equity Focused and Trauma-Informed Communication Intervention — Clinician communication intervention that includes didactic training and real-time feedback on communication behaviors during clinical encounters.

SUMMARY:
Development and pilot testing of a clinician coaching communication intervention to improve communication between medical teams and caregivers (parents, family members) of children in the hospital. Our team is specifically focused on improving partnership, respect, and collaboration with Black and Latinx caregivers of children in the hospital by incorporating elements from trauma-informed care and racial equity into a communication intervention. The investigators will explore the impact of this intervention on communication quality, caregiver trust, caregiver satisfaction, and hospital readmissions.

DETAILED DESCRIPTION:
When admitted to the hospital, Black and Latino(a/x) children are at greater risk of medical errors, surgical complications, longer, more-costly hospital stays, and mortality compared to White children. Although many factors play a role, poor clinician communication likely contributes to these disparities in health outcomes. Across settings, including our preliminary work in the inpatient pediatric environment, Black and Latino(a/x) patients have been shown to experience worse communication quality as evidenced by less patient and family-centered, empathic, and respectful communication as compared to White patients. Poor communication can make the hospital stay more stressful for caregivers, with implications for caregiver and child health and recovery from illness. While prior experiences of discrimination and trauma can negatively affect clinician-caregiver communication, current best practices in clinician communication fail to incorporate equity and trauma-informed principles. In this study the investigators will test the feasibility, acceptability, and preliminary efficacy of a pilot randomized waitlist control trial of an equity focused and trauma-informed clinician coaching communication intervention that aims to teach clinicians skills to improve communication in areas where inequities are known to exist (i.e. respect, partnership) and incorporate principles of equity (i.e affirmation) and trauma-informed care. To do this, first the investigators will co-develop and refine a clinician coaching communication intervention with iterative feedback from Black and Latino(a/x) caregivers as well as clinicians of children in the hospital. Second, the investigators will examine the feasibility, acceptability and preliminary efficacy of the intervention. The investigators will randomize 10 clinicians to an intervention or waitlist group; clinicians in the intervention group will receive the intervention immediately, while clinicians in the waitlist group will initially serve as the control arm then receive the intervention to provide feasibility and acceptability data. The investigators will assess the feasibility of recruiting and collecting data as well as acceptability of the intervention by clinicians. The investigators will explore preliminary efficacy for the effect of the intervention on communication, caregiver satisfaction, caregiver trust, and hospital readmissions.

ELIGIBILITY:
Eligibility criteria for caregivers:

* Adults (18 years of age or older)
* Proficient in English or Spanish
* Capable of providing informed consent
* Identified as a primary caregiver (parent or guardian) of a hospitalized Black or Latino(a/x) child on the general pediatrics team.
* We will exclude caregivers of children undergoing evaluation for child abuse/neglect or other cases in which the medical team believes family-centered rounds are not appropriate.

Eligibility criteria for clinicians:

* pediatric attending physicians who provide hospital care to children at Duke Children's Hospital.
* Capable of providing informed consent
* We will exclude clinicians who do not provide hospital care to children on the general pediatrics team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-03-29 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by enrollment rate of clinicians and caregivers combined | Up to 12 months
Feasibility measured by the rate of complete data collection by caregivers | Up to 12 months
Fidelity measured by the rate of intervention elements completed per encounter by clinicians | Up to 12 months
Acceptability of the intervention as measured by the Acceptability of Intervention Measure (AIM) | Up to 12 months
  The AIM has 4 items. Each with response of 5 point likert scale (completely disagree to completely agree). The Investigator will assign a score of 1 to completely disagree and a 5 to completely agree for each item. To calculate the AIM the Investigator average together the responses to the 4 items.
Appropriateness measured by the Intervention Appropriateness Measure (IAM) | Up to 12 months
  The IAM has 4 items. Each with response of 5 point likert scale (completely disagree to completely agree). The Investigator will assign a score of 1 to completely disagree and a 5 to completely agree for each item. To calculate the AIM the Investigator average together the responses to the 4 items.
Feasibility measured by the Feasibility of Intervention Measure (FIM) | Up to 12 months
  The FIM has 4 items. Each with response of 5 point likert scale (completely disagree to completely agree). The Investigator will assign a score of 1 to completely disagree and a 5 to completely agree for each item. To calculate the AIM the Investigator average together the responses to the 4 items.
Number of Clinician rapport-building statements | Up to 12 months
  Clinician communication behaviors measured via audio-recorded hospital encounters.
Number of Clinician partnership-building statements | Up to 12 months
  Clinician communication behaviors measured via audio-recorded hospital encounters.
Number of Clinician interruptions | Up to 12 months
  Clinician communication behaviors measured via audio-recorded hospital encounters.
Number of Clinician praise statements | Up to 12 months
  Clinician communication behaviors measured via audio-recorded hospital encounters.
Number of Clinician permission asking | Up to 12 months
  Clinician communication behaviors measured via audio-recorded hospital encounters.
Caregiver Satisfaction measured by survey | Up to 12 months
  1 item question on the post-rounds caregiver survey. Response choices will include: not at all satisfied, a little satisfied, satisfied, and extremely satisfied.
Caregiver Trust in their Childs Doctors measured by the Wake Forest Physician Trust Scale | Up to 12 months
  The Wake Forest Physician Trust Scale is a validated 5 item instrument on the post-rounds caregiver survey. Responses to the 5 items are summed together and can vary from a score of 5-25. A higher score indicates a more positive outcome.
Caregiver Reported Communication Quality measured by the Interpersonal Processes of Care Short Form | Up to 12 months
  The interpersonal processes of care measure has 18 items on the short form, each with response of Never (score=1), Rarely (Score=2), Sometimes (Score=3), Usually (Score=4), Always(Score=5). The Investigator will average together responses from the 18 items to give a value from 1-5 for each domain.
Caregiver Stress | Timeframe up to 12 months
  Measured by salivary cortisol levels

SECONDARY OUTCOMES:
Number of Caregiver Participatory Behaviors | Up to 12 months
  The investigators will measure caregiver participation during clinical encounters by counting the number of times caregivers (1) ask a question, (2) state a preference and (3) express an emotion per clinician encounter. These three behaviors will be summed together and analyzed in aggregate as a count of caregiver participatory behaviors.
Number of participants with Hospital Readmission at 30 days | 30 days after discharge
  Child unplanned hospital readmission
Number of participants with Hospital Readmission at 90 days | 90 days after discharge
  Child unplanned hospital readmission
Caregiver ability to correctly identify child's diagnosis | Up to 12 months
  Using validated approach described by Lion et al. the caregiver description of "the main condition child was admitted for" will be compared to the diagnoses listed by the child's doctors in the electronic health record.
Change in caregiver Salivary Cortisol | 30-60 minutes before and 20-30 minutes after FCR
  The investigators will assess for reductions in caregiver salivary cortisol following interactions with clinical teams. The investigators will collect saliva samples from caregivers at two time points: 30-60 minutes before and 20-30 minutes after family-centered rounds (FCR). The investigators anticipate lower salivary cortisol levels in the intervention compared to control arm at 20-30 minutes following FCR. The investigators will also compare differences in the change in cortisol from before and after FCR for each caregiver; the investigators hypothesize caregivers in the intervention arm will have a smaller change from baseline following FCR.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M. Parente, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Sustem, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be available to individuals on the Institutional Review Board protocol. We will share study protocol documents including intervention didactic materials and outcome measure assessments.

REFERENCES:
- [Background] Parente VM, Khan A, Robles JM. Belonging on Rounds: Translating Research Into Inclusive Practices for Families With Limited English Proficiency to Promote Safety, Equity, and Quality. Hosp Pediatr. 2022 May 1;12(5):e171-e173. doi: 10.1542/hpeds.2022-006581. No abstract available. PMID 35411380
- [Result] Khan A, Parente V, Baird JD, Patel SJ, Cray S, Graham DA, Halley M, Johnson T, Knoebel E, Lewis KD, Liss I, Romano EM, Trivedi S, Spector ND, Landrigan CP; Patient and Family Centered I-PASS SCORE Scientific Oversight Committee; Bass EJ, Calaman S, Fegley AE, Knighton AJ, O'Toole JK, Sectish TC, Srivastava R, Starmer AJ, West DC. Association of Patient and Family Reports of Hospital Safety Climate With Language Proficiency in the US. JAMA Pediatr. 2022 Aug 1;176(8):776-786. doi: 10.1001/jamapediatrics.2022.1831. PMID 35696195
- [Result] Parente V, Stark A, Key-Solle M, Olsen M, Sanders LL, Bartlett KW, Pollak KI. Caregiver Inclusivity and Empowerment During Family-Centered Rounds. Hosp Pediatr. 2022 Feb 1;12(2):e72-e77. doi: 10.1542/hpeds.2021-006034. PMID 35079809

DOCUMENTS (1):
  • Informed Consent Form (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT05618652/ICF_000.pdf